CLINICAL TRIAL: NCT00324389
Title: A Pilot Study to Characterize Interferon-Induced Gene Expression in Liver Cells and Peripheral Blood Lymphocytes Using High Density Oligonucleotide Microarray Expression Analysis in Caucasian and African American Patients With Chronic Hepatitis C
Brief Title: Interferon-Induced Gene Expression in Liver Cells and Peripheral Blood Lymphocytes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-014
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2009-04

CONDITIONS: Hepatitis C
Keywords: Interferon, Gene Expression in Liver, Lymphocytes, High Density Oligonucleotide Microarray Expression Analysis, African American, Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Interferon-alpha

INTERVENTIONS:
Drug: Interferon alpha

SUMMARY:
This proposal seeks to use DNA analyses to understand how racial and genetic factors influence interferon (treatment) response in HCV infection in African Americans. A better understanding should allow rational design of new therapies or better use of existing therapies. Patients will provide medical history and undergo a physical exam, blood draws, electrocardiogram, possible chest x-ray, and abdominal ultrasound. Patients will be admitted to the hospital for 5 days and undergo 2 liver biopsies, sedation, and multiple blood draws. Twenty adult male volunteers (10 Caucasians,10 African Americans) ages 18 - 65 years will participate.

DETAILED DESCRIPTION:
This proposal uses sophisticated DNA microarray analyses of the transcriptional changes induced in hepatocytes (cellular locus of viral replication) and peripheral blood lymphocytes (one compartment of immune responder cells) in an effort to better understand how racial and host genetic factors influence interferon response in HCV infection. A better understanding of these underlying mechanisms should allow rational design of new therapies or better use of existing therapeutic modalities. The variables to be investigated are racial differences in interferon induced: 1) HCV viral kinetics and 2) intrahepatic and PBL transcriptional responses. Specific Aim 1: (a) To compare the phase 1 and early phase 2 decline of the viral titer in serum in African-Americans and Caucasians following a single dose of IFN-alpha (10 MU sc). (b) To determine the hepatic HCV RNA abundance in both a baseline liver biopsy and in a repeat liver biopsy taken 24 hrs after administration of interferon, and to determine how this correlates with the HCV RNA decline in serum over the 24 hr period. (c) To compare the rates of viral decline in the liver and serum in African-Americans and Caucasians 24 hours after interferon, and to relate this to the pharmacokinetics (PK) of the initial dose of interferon. A total of 10 Caucasian and 10 African American patients with chronic hepatitis C and HCV genotype 1 will be enrolled in this study. All study patients will undergo a baseline percutaneous liver biopsy on day 1 of the study. On day 3, a single dose of IFN-alpha 2a (10 MU sc) will be administered and a repeat liver biopsy will be done 24 hours after the injection. Specific Aim 2: (a) To utilize Affymetrix HG-U133A&B Human GeneChips® to determine global mRNA profiles in liver tissue collected from patients before and 24 hrs after a single 10 MU dose of IFN-alpha and thereby assess the intrahepatic transcriptional response to IFN-alpha. (b) To characterize differences in the early intrahepatic transcriptional response to interferon in Caucasians and African Americans. Specific Aim 3: (a) To utilize Affymetrix HG-U133A&B Human GeneChips® to determine global transcription profiles in peripheral blood lymphocytes pre-treatment, 24hrs, and 48hrs after the initial dose of interferon and to compare these results in Caucasians and African Americans at these time points. (b) To compare global gene profiles in lymphocytes and liver at baseline and 24hrs after interferon, and determine whether lymphocytic transcriptional profiling is a valid surrogate for intrahepatic gene profiling. Specific Aim 4: To use sophisticated bioinformatics approaches and HCV kinetic modeling to determine whether differences in early intrahepatic or lymphocytic transcriptional profiles correlate with early changes in the level of viremia (observed antiviral response) in the period immediately following administration of the 10 MU dose of IFN-alpha.

ELIGIBILITY:
Inclusion Criteria:

1. Male non-Hispanic African-American or non-Hispanic Caucasian patients between 18 and 65 years of age
2. Abstinence from any ingestion of alcohol and smoking for at least 7 days prior to study for those who drink or smoke socially
3. HCV genotype 1 (1a, 1b or mixture of 1a and 1b). HCV genotyping will be performed at the Molecular Diagnostic Laboratory at UTMB using the LiPA assay (Innogenetics)
4. Presence of HCV RNA in serum (>10 [to the fifth power] copies/ml)
5. Not previously treated with any interferon and/ or ribavirin
6. Compensated liver disease with the following laboratory criteria:

   * Hemoglobin greater than or equal to 13 gm/dl for males
   * Granulocyte count greater than or equal to 1,000/cubic mm
   * Platelets greater than or equal to 100,000/cubic mm
   * Prothrombin time <2 sec. elevation
   * Total bilirubin (0.1-1.1 mg/dl). If elevated, the conjugated Bilirubin must be within normal limits (0-0.3 mg/dl)
   * Serum albumin within normal limits (3.5-5.0 g/dl)
   * Serum creatinine within normal limits (0.7-1.7 mg/ml)
7. Absence of other known causes of liver disease (e.g. autoimmune hepatitis, hemochromatosis, Wilson's diseases, alpha-1 anti-trypsin deficiency, drug-induced liver injury, alcoholic liver disease)
8. No other systemic antiviral or immunosuppressive therapy within the last 6 months
9. Absence of concurrent medical and psychiatric illnesses (e.g. other viral co-infection such as HBV or HIV, renal failure, poorly controlled diabetes, cardiac-pulmonary diseases, CNS disease, active alcoholism, depression, psychosis)
10. No history of Type 1 or Type 2 diabetes mellitis
11. TSH within normal limits (0.49-4.7 micro IU/ml)
12. ANA <1:160
13. No history of hepatocellular carcinoma
14. Alpha fetoprotein within normal limits (0-20 ng/ml) obtained within 6 months of enrollment.
15. If participating in sexual activity that could lead to pregnancy, the study volunteer must agree that two reliable methods of contraception will be used with his partner simultaneously while receiving medication, and for 6 months after stopping the medications. The following are considered reliable and effective methods of birth control.

1) Condoms with or without a spermicidal agent 2) Diaphragm or cervical cap with spermicide 3) IUD 4) Hormonal-based contraception 16. Exceptions may include if study participant/partner is surgically sterile 17. Willingness to comply with procedures and treatment as outlined in the protocols and provide written informed consent

Exclusion Criteria:

1. Interferon or ribavirin therapy at any previous time
2. Any investigational drug <= 24 weeks prior to the first dose of study drug
3. Any alternative or folk medicine within 24 weeks of screening
4. Any systemic antiviral therapy <= 24 weeks prior to the first dose of study drug or expectation that such treatment will be needed at any time during the study. Exception: patients who have taken or are expected to require acyclovir for herpetic lesions
5. Patient with a baseline increased risk for anemia (e.g. hemoglobinopathies such as thalassemia, spherocytosis, sickle cell anemia or a history of symptomatic recurring GI bleeding, etc.) or for whom anemia would be medically problematic
6. Evidence of alcohol and/or drug abuse within 6 months
7. History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, clinical evidence of rheumatoid arthritis)
8. Evidence of an active or suspected cancer or a history of malignancy
9. History of having received any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) <= 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study
10. History of major organ transplantation with an existing functional graft
11. History of bone marrow transplantation
12. Anything that in the opinion of the investigator puts the patient at increased risk, or increases the likelihood that the patient may not be able to complete the protocol

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2
Dates: Start 2006-05; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States